CLINICAL TRIAL: NCT01611155
Title: A Pilot Randomized, Placebo-controlled, Double Blind Study of Venlafaxine to Prevent Oxaliplatin-Induced Neuropathy
Brief Title: Venlafaxine in Preventing Chronic Oxaliplatin-Induced Neuropathy In Patients Receiving Combination Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC11C4; NCI-2012-00318 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2018-10

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (management of therapy complications) (Experimental): Patients receive venlafaxine PO BID beginning on day 1 of and continuing through completion of FOLFOX.
  Interventions: Drug: venlafaxine; Other: questionnaire administration; Other: quality-of-life assessment
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID beginning on day 1 of and continuing through completion of FOLFOX.
  Interventions: Drug: placebo; Other: questionnaire administration; Other: quality-of-life assessment

INTERVENTIONS:
Drug: venlafaxine — Given PO
  Other Names: Effexor; VNF
  Arms: Arm I (management of therapy complications)
Drug: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: questionnaire administration — Ancillary studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
You are being asked to take part in this research study because you are going to be treated with oxaliplatin chemotherapy as part of your standard care. Oxaliplatin commonly causes neuropathy (numbing, tingling and/or pain).The purpose of this study is to compare the effects, good and/or bad, of venlafaxine with a placebo (an inactive agent) on oxaliplatin-induced neuropathy (numbing, tingling and/or pain)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore whether venlafaxine can prevent or ameliorate chronic, cumulative neurotoxicity associated with oxaliplatin in cancer patients receiving oxaliplatin, fluorouracil, leucovorin calcium (FOLFOX).

SECONDARY OBJECTIVES:

I. To explore whether venlafaxine can ameliorate acute neuropathy associated with oxaliplatin.

TERTIARY OBJECTIVES:

I. To explore whether venlafaxine can increase the cumulative oxaliplatin doses that can be delivered without dose-limiting chronic neurotoxicity.

II. To explore whether venlafaxine causes adverse events in this setting. III. To explore whether the neuropathy data provided by the Rydel-Seiffer graduated tuning fork is consistent with patient-reported outcome (PRO) measures of chemotherapy-induced peripheral neuropathy (CIPN) and whether this tool might cause different results in patients receiving venlafaxine versus placebo.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive venlafaxine orally (PO) twice daily (BID) beginning on day 1 of and continuing through completion of FOLFOX.

ARM II: Patients receive placebo PO BID beginning on day 1 of and continuing through completion of FOLFOX.

After completion of study treatment, patients are followed up at 1, 3, 6, 12, and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive FOLFOX chemotherapy with individual oxaliplatin doses of 85 mg/m^2 per cycle given in 2 week cycles (e.g. modified [m] FOLFOX6 or FOLFOX4) Adequate complete blood count (CBC) and creatinine values (per attending physician) obtained =< 28 days prior to registration Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0, 1 or 2 Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential Ability to complete questionnaire(s) by themselves or with assistance Life expectancy >= 4 months Strong inhibitors of CYP3A4: > 5-fold increase in the plasma area under the curve (AUC) values or more than 80 % decrease in clearance

  * Indinavir (Crixivan®)
  * Nelfinavir (Viracept®)
  * Atazanavir (Reyataz®)
  * Ritonavir (Norvir®)
  * Clarithromycin (Biaxin®, Biaxin XL®)
  * Itraconazole (Sporanox®)
  * Ketoconazole (Nizoral®)
  * Nefazodone (Serzone®)
  * Saquinavir (Fortovase®, Invirase®)
  * Telithromycin (Ketek®) Inducers of CYP3A4
  * Efavirenz (Sustiva®)
  * Nevirapine (Viramune®)
  * Carbamazepine (Carbatrol®, Epitol®, Equetro™, Tegretol®, Tegretol-XR®)
  * Modafinil (Provigil®)
  * Phenobarbital (Luminal®)
  * Phenytoin (Dilantin®, Phenytek®)
  * Pioglitazone (Actos®)
  * Rifabutin (Mycobutin®)
  * Rifampin (Rifadin®)
  * St. John's wort

Exclusion Criteria:

Any of the following:

* Pregnant women
* Nursing women History of an allergic reaction to, or intolerance of, venlafaxine Treatment =< 7 days with other antidepressants, anticonvulsants, monoamine oxidase (MAO) inhibitors, or other neuropathic pain medication agents such as carbamazepine, phenytoin, valproic acid, gabapentin, lamotrigine, topical lidocaine patch or gel, capsaicin cream, or amifostine; in addition, they may not be taking other agents for the treatment of neuropathy, nor other known moderate or strong CYP 2D6 (which consist of Cinacalcet [Sensipar™], quinidine, and Terbinafine [Lamisil®, Lamisil AT®]), nor the strong inducer of CYP 2D6 terbinafine (Lamisil®, Lamisil AT®), nor the following drugs that substantially effect CYP 3A4 Moderate inhibitors of CYP3A4: > 2-fold increase in the plasma AUC values or 50-80% decrease in clearance
* Aprepitant (Emend®)
* Erythromycin (Erythrocin®, E.E.S. ®, Ery-Tab®, Eryc®, EryPed®, PCE®
* Fluconazole (Diflucan®)
* Grapefruit juice
* Verapamil (Calan®, Calan SR®, Covera-HS®, Isoptin SR®, Verelan®, Verelan PM®)
* Diltiazem (Cardizem®, Cardizem CD®, Cardizem LA®, Cardizem SR®, Cartia XT™, Dilacor XR®, Diltia XT®, Taztia XT™, Tiazac®) Other medical conditions which, in the opinion of the treating physician/allied health professional, would make this protocol unreasonably hazardous for the patient Prior neurotoxic chemotherapy Concurrent radiotherapy Current (within the last month) pre-existing peripheral neuropathy of any grade Uncontrolled hypertension (defined as 3 consecutive readings over the past year of over 160 systolic, and over 100 diastolic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02-17 (Actual); Primary Completion 2014-03-07 (Actual); Study Completion 2015-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Zimmerman C, Atherton PJ, Pachman D, Seisler D, Wagner-Johnston N, Dakhil S, Lafky JM, Qin R, Grothey A, Loprinzi CL. MC11C4: a pilot randomized, placebo-controlled, double-blind study of venlafaxine to prevent oxaliplatin-induced neuropathy. Support Care Cancer. 2016 Mar;24(3):1071-8. doi: 10.1007/s00520-015-2876-5. Epub 2015 Aug 8. PMID 26248652

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Venlafaxine): Patients receive venlafaxine PO BID beginning on day 1 of and continuing through completion of FOLFOX.
Period: Overall Study
Arm/Group | Arm I (Venlafaxine) | Arm II (Placebo)
Started | 25 | 25
Received Treatment | 25 | 25
Completed (Evaluable for primary endpoint) | 16 | 18
Not Completed | 9 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Refused further treatment | 6 | 4
Not completed — Disease progression | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Alternative treatment | 0 | 1
Not completed — Ineligible patient | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients summarized in the baseline characteristics table exclude ineligible and patient withdrawals.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Venlafaxine) | Arm II (Placebo) | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (11.3) | 58.4 (10.3) | 60.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Cycle 1 Sensory Neuropathy Score (Items 31-36, 39, 40 and 48) of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-CIPN20
Description: The EORTC QLQ-CIPN20 sensory neuropathy score will be calculated using the standard algorithm of EORTC QLQ-CIPN20 and transformed into a 0-100 point scale, where high scores meant less symptom burden. The changes of sensory neuropathy from baseline will be derived by subtracting the baseline score from the sensory neuropathy scores at each cycle of evaluation.
Time Frame: Up to 2 weeks
Population: Patients who completed the (QLQ)-CIPN20 Sensory neuropathy items at cycle 1 are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Venlafaxine) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 20
score on a scale | 96.22 (5.88) | 95.83 (8.84)
Statistical Analysis 1: Comparison: Arm I (Venlafaxine) vs Arm II (Placebo); Test type: Superiority; p = 0.87, t-test, 2 sided

2. Secondary Outcome: Cycle 1 Acute Neuropathy as Measured by EORTC QLQ CIPN20 Motor Subscale (Items 37, 38, 41-45 and 49), and Autonomic Scale (Items 46, 47, 50)
Description: The EORTC QLQ-CIPN20 motor and autonomic neuropathy scores will be calculated using the standard algorithm of EORTC QLQ-CIPN20 and transformed into a 0-100 point scale, where high scores meant less symptom burden. The changes of sensory neuropathy from baseline will be derived by subtracting the baseline score from the sensory neuropathy scores at each cycle of evaluation.
Time Frame: Up to 2 weeks
Population: There were a few Venlafaxine patients who completed the items for the motor subscale but did not complete the items for autonomic subscale in cycle 1 and thus the number analyzed for each subscale is different on the venlafaxine arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Venlafaxine) | Arm II (Placebo)
Number analyzed (Participants) | 20 | 21
score on a scale
  Motor subscale | 97.28 (6.33) | 95.98 (6.82)
  Autonomic subscale: number analyzed (Participants) | 18 | 21
  Autonomic subscale | 91.36 (15.03) | 90.74 (12.34)
Statistical Analysis 1: Comparison: Arm I (Venlafaxine) vs Arm II (Placebo); Motor subscale; Test type: Superiority; p = 0.53, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm I (Venlafaxine) vs Arm II (Placebo); autonomic subscale; Test type: Superiority; p = 0.89, t-test, 2 sided

ADVERSE EVENTS:
Description: All patients who received treatment and submitted an AE form are included in the summary below.
Arm/Group | Arm I (Venlafaxine) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 1/24 | 1/25
Serious Adverse Events (participants affected / at risk) | 2/24 | 2/25
Other Adverse Events (participants affected / at risk) | 21/24 | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Venlafaxine) (N=24) | Arm II (Placebo) (N=25)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Venlafaxine) (N=24) | Arm II (Placebo) (N=25)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 15 (52) | 14 (47)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (3) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (19) | 4 (7)
Platelet count decreased (Investigations) | 1 (7) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (3)
Somnolence (Nervous system disorders) | 4 (4) | 2 (17)
Agitation (Psychiatric disorders) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 5 (19) | 1 (1)
Hypertension (Vascular disorders) | 7 (34) | 10 (57)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes